CLINICAL TRIAL: NCT06146270
Title: National Register of Postoperative Outcomes in the Russian Federation: a Multicenter Observational Study
Brief Title: Russian Registry of Surgical OutcomeS
Acronym: RuSOS
Status: Recruiting | Type: Observational
Sponsor: Russian Federation of Anesthesiologists and Reanimatologists (Other)
Collaborators: Kuban State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: FARCT0005
Record Dates: First submitted 2023-11-18; First posted 2023-11-24 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Surgery; Anesthesia; Outcome, Fatal; Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: A cohort in which the incidence of the primary outcomes in the study population will be assessed.
- Cohort B: A cohort in which risk factors for primary outcomes will be identified, and a risk calculator for their development will be developed and validated

SUMMARY:
Identification of risk factors that cause a high probability of an unfavorable outcome in the postoperative period is an urgent problem. The creation of national databases (registries) makes it possible to maximally cover a certain patient population by identifying its characteristic risk predictors. As literature data show, existing registries differ in the criteria for inclusion in the study, in the characteristics of the populations studied, and there is often no common view on the classification of postoperative outcomes. Goal of a study is a creation of a Russian national calculator for the risk of postoperative complications and mortality.

Two-level observational retrospective-prospective study was planned. Setting: National multicenter study of surgical inpatients. Patients: Adult patients undergoing elective and emergency surgery. Types of interventions: in obstetrics, in gynecology, on the breast, in urology and kidneys, in endocrine surgery, in maxillofacial surgery, in orthopedics and traumatology, on the lower floor of the abdominal cavity, on the liver and biliary tract, on the upper floor of the abdominal cavity cavities, in thoracic surgery, in vascular surgery, in neurosurgery, in cardiac surgery, in other areas (with mandatory specification).

The study was organized by the Federation of Anesthesiologists and Reanimatologists of Russia. Primary (30-day mortality, 30-day complications) and secondary (hospital mortality, hospital complications, length of stay in anesthesiology, resuscitation and intensive care departments, length of hospital stay, multiple organ failure (2 or more points on the SOFA scale (Sequential)) Organ Failure Assessment), 90-day mortality, 90-day complications, intensive care after-effects syndrome, readmission, 1-year mortality) outcomes were determined. The required sample size and statistical analysis methods are described. The planned duration of the study is 2024-2028.

DETAILED DESCRIPTION:
Currently, the incidence of perioperative complications and mortality associated with surgical intervention are minimized. However, taking into account the significant number of surgical interventions performed worldwide (more than 300 million per year), the total number of patients with complicated postoperative periods is large, and postoperative mortality ranks third in the structure of causes of death (7, 7%), second only to coronary heart disease and stroke. Moreover, even in discharged patients, complications that develop can significantly reduce quality of life and worsen long-term prognosis. To a greater extent, the above applies to high-risk patients, whose identification is a priority task of anesthesiology.

Identification of risk factors that cause a high probability of an unfavorable outcome is currently unthinkable without conducting comprehensive prospective population-based studies, which, on the one hand, make it possible to assess the contribution of many variables to the risk of complications and mortality, and on the other hand, to maximally cover a certain population by identifying characteristic predictors for it. To date, several population-based studies and programs have been described in the literature that have led to the creation of national databases (registries) of postoperative outcomes. Such studies include several international (ISOS, EuSOS and ASOS) and national ones, such as SweSOS [8] or ColSOS , which are at different stages of implementation. Among the national databases, the best known is the ACS-NSQIP (American College of Surgeons National Surgical Quality Improvement Program) database, which contains information on the outcomes of surgical treatment for more than 5 million patients in the United States since 1991 .

The results obtained from these studies often vary widely, due to the diversity of approaches to study inclusion criteria, differences in the characteristics of the populations studied, and the lack of a uniform view on the classification of postoperative outcomes. When assessing mortality, the authors most often record 30-day mortality, however, taking into account modern ideas about the role of perioperative factors and complications in the development of an unfavorable long-term outcome, the need to determine one-year mortality becomes obvious. As shown by the national observational study SweSOS, the mortality rate increases significantly over time, with 30-day mortality being 1.8%, 3-month mortality - 3.9%, and 6-month and annual mortality - 5.0% and 8.5% , respectively .

There is also no uniform approach to the registration of postoperative complications, and modern protocols use several systems, the most common of which are the classification of the joint working group of ESA (The European Society of Anesthesiologists) and ESICM (The European Society of Intensive Care Medicine, The European). Society of Intensive Care Medicine) and the ACS-NSQIP classification (The American College of Surgeons (ACS) National Surgical Quality Improvement Program (NSQIP)). And although they are similar in many ways (complications are grouped into blocks according to the nature of the disorders), differences are also present, and even the same complication may have a different definition. In addition, some significant outcomes are not included in these classifications, which predetermines their underestimation.

Of course, one of the advantages of creating a large population-based database is the recording of a large number of potential predictors of adverse outcome and subsequent assessment of their individual contribution to the complex perioperative risk. The type of surgical intervention itself is a factor that largely determines the likelihood of complications.

The goal is to create a Russian national calculator for the risk of postoperative complications and mortality.

Primary target points:

1. Creation of a national register of postoperative outcomes in different areas of surgery.
2. Determination of the frequency and structure of outcomes after elective and emergency surgery.
3. Identification of predictors of unfavorable outcome.
4. Development and validation of a model for predicting complications and mortality in various areas of surgery
5. Creation of calculators for the risk of postoperative complications and mortality in various fields of surgery and their integration into a single calculator
6. Analysis of long-term results in patients with postoperative complications (90 days and a year after surgery)

Secondary target points:

1. The role of concomitant diseases in the development of unfavorable outcome
2. The influence of age on primary and secondary postoperative outcomes
3. The influence of the type of anesthesia on the course of the postoperative period
4. The influence of oncological pathology and specific treatment on primary and secondary postoperative outcomes
5. The impact of the urgency of surgery on the risk of an unfavorable outcome
6. Influence of localization, access and duration of surgery on postoperative outcome
7. Assessment and validation of surgical and anesthesiological risk scales for lethal outcome (can be listed)
8. Evaluation and validation of surgical and anesthetic risk scales for primary and secondary outcomes
9. Stratification of patients at high perioperative risk with details on cardiac, respiratory, neurological, renal, hepatic, hemostasiological, infectious and others.
10. Influence of quality criteria for implementation of FAR recommendations on the course of the postoperative period
11. Analysis of the course of ICU-syndrome in patients with complications and depending on the maximum score on the SOFA scale and the structure of MOF in the postoperative period
12. Analysis of the effectiveness of rehabilitation measures in patients with ICU-syndrome
13. Analysis of the causes of mortality (based on autopsy reports and clinical and laboratory data of patients).

Cohort A

The checklist (basic) is filled out for all patients with postoperative complications. At the same time, the total number of patients operated on in a particular center is taken into account on a quarterly basis, taking into account their distribution by area of surgery. Based on the data from the basic checklist, answers will be received to the following target points:

1. Creation of a national register of postoperative outcomes in different areas of surgery.
2. Determination of the frequency and structure of outcomes after planned and emergency surgical interventions.
3. Analysis of long-term results in patients with postoperative complications (90 days and a year after surgery)
4. Analysis of the course of ICU-syndrome in patients with complications and depending on the maximum score on the scale and the structure of MOF in the postoperative period
5. Analysis of the effectiveness of rehabilitation measures in patients with ICU syndrome

Cohort B Basic checklist plus additional checklist: completed for all operated patients within one selected week quarterly The total number of patients operated on in a particular center is also taken into account quarterly, taking into account their distribution by area of surgery.

Based on the data from the basic and additional checklists, answers to the most important target points (3 primary and 10 secondary) will be obtained:

1. Identification of predictors of unfavorable outcome.
2. Development and validation of a model for predicting complications and mortality in various fields of surgery
3. Creation of calculators for the risk of postoperative complications and mortality in various fields of surgery and their integration into a single calculator
4. The role of concomitant diseases in the development of unfavorable outcome
5. The influence of age on primary and secondary postoperative outcomes
6. The influence of the type of anesthesia on the course of the postoperative period
7. The influence of oncological pathology and specific treatment on primary and secondary postoperative outcomes
8. The impact of the urgency of surgery on the risk of an unfavorable outcome
9. The influence of localization, access and duration of surgery on postoperative outcome
10. Assessment and validation of surgical and anesthesiological risk scales for lethal outcome (can be listed)
11. Evaluation and validation of surgical and anesthetic risk scales for primary and secondary outcomes
12. Stratification of patients at high perioperative risk with details on cardiac, respiratory, neurological, renal, hepatic, hemostasiological, infectious and others.
13. Influence of quality criteria for implementation of FAR recommendations on the course of the postoperative period

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 years and older) undergoing elective surgery:

  * In obstetrics
  * In gynecology
  * Breast
  * In urology and kidneys
  * In endocrine surgery
  * In maxillofacial surgery
  * In orthopedics and traumatology
  * On the lower abdominal cavity
  * On the liver and biliary tract
  * On the upper abdominal cavity
  * In thoracic surgery
  * In vascular surgery
  * In neurosurgery
  * In cardiac surgery
  * In other areas (with mandatory specification)
* Adult patients (age 18 years and older) undergoing emergency surgery in the listed and other areas of surgery (for example, in purulent surgery).

Exclusion Criteria:

1. Lack of informed consent from the patient
2. Complications associated with the manipulations of an anesthesiologist
3. Interventions without the participation of an anesthesiologist-resuscitator
4. Incomplete checklists
5. Errors when filling checklists
6. Deviations from the Register protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing surgery in various areas of surgery
Sampling Method: Probability Sample
Enrollment: 162000 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative mortality | up to 30 days after surgery
  Incidence of postoperative death defined as any death occurring during and up to 30 days after surgery
Postoperative complications | up to 30 days after surgery
  Incidence of the following complications with severity due to Clavien-Dindo classification:
  Arrhythmia Cardiac arrest Cardiogenic pulmonary edema Deep vein thrombosis Myocardial infarction Myocardial damage after non-cardiac operations Pulmonary embolism Postoperative transfusion Postoperative delirium Stroke ARDS Acute respiratory failure Pneumonia Pleural effusion Atelectasis Respiratory infection Bronchospasm Pneumothorax Aspiration pneumonitis Reintubation Renal injury Infection without a specific source Laboratory confirmed bacteremia Superficial wound infection Deep wound infection Postoperative infection Urinary tract infection Sepsis Septic shock Gastrointestinal bleeding Paralytic ileus Postoperative bleeding Anastomotic leakage Dehiscence of wound Other Malignant hyperthermia Anaphylaxis Anaphylactic shock Fat embolism

SECONDARY OUTCOMES:
Length of stay in the ICU | up to 30 days after surgery
  Number of days in the ICU
Length of hospital stay | up to 30 days after surgery
  Number of days in the hospital
Multiple organ failure (2 or more points on the SOFA (Sequential Organ Failure Assessment) scale) | up to 30 days after surgery
  Incidence of MOF
90-days mortality | up to 90 days after surgery
  Incidence of postoperative death defined as any death occurring during and up to 90 days after anaesthesia
90-days postoperative complications | up to 90 days after surgery
  Incidence of the following complications with severity due to Clavien-Dindo classification:
  Arrhythmia Cardiac arrest Cardiogenic pulmonary edema Deep vein thrombosis Myocardial infarction Myocardial damage after non-cardiac operations PE Postoperative transfusion Postoperative delirium Stroke ARDS Acute respiratory failure Pneumonia Pleural effusion Atelectasis Respiratory infection Bronchospasm Pneumothorax Aspiration pneumonitis Reintubation Renal injury Infection without a specific source Laboratory confirmed bacteremia Superficial wound infection Deep wound infection Postoperative infection Urinary tract infection Sepsis Septic shock Gastrointestinal bleeding Paralytic ileus Postoperative bleeding Anastomotic leakage Dehiscence of wound Other Malignant hyperthermia Anaphylaxis Anaphylactic shock Fat embolism
ICU - syndrome | up to 90 days after surgery
  The intensive care unit (ICU) syndrome is a type of organic brain syndrome manifested by a variety of psychological reactions, including fear, anxiety, depression, hallucinations, and delirium.
Readmission | up to 1 year after surgery
  Any readmission to the hospital
1-year mortality | up to 1 year after surgery
  Incidence of death defined as any death occurring during and up to 1 year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Igor Zabolotskikh, MD, Study Chair — Kuban State Medical University; Nikita Trembach, MD, Study Director — Kuban State Medical University; Andrey Belkin, MD, Study Director — Clinical Institute of Brain; Evgeniy Grigiriev, MD, Study Director — Research Institute for Complex Issues of Cardiovascular Diseases; Alexei Gritsan, MD, Study Director — Voino-Yasenetsky Krasnoyarsk State Medical University; Pavel Dunts, PhD, Study Director — Pacific State Medical University; Vadim Ershov, MD, Study Director — Orenburg State Medical University; Mikhail Kirov, MD, Study Director — Northern State Medical University; Artem Kuzovlev, MD, Study Director — Federal Research and Clinical Center of Intensive Care Medicine and Rehabilitology; Alexandr Kulikov, MD, Study Director — Ural State Medical University; Alexey Ovezov, MD, Study Director — Moscow Regional Research and Clinical Institute; Denis Protsenko, MD, Study Director — Pirogov Russian National Research Medical University; Valeriy Subbotin, MD, Study Director — Loginov Moscow Clinical Scientific Center; Victoria Khoronenko, MD, Study Director — P. A. Hertsen Moscow Oncology Research Center; Efim Shifman, MD, Study Director — Moscow Regional Research and Clinical Institute, Moscow, Russia; Alexey Shchegolev, MD, Study Director — Military Medical Academy, Bulgaria; Konstantin Lebedinskii, MD, Study Director — North-Western State Medical University named after Ilya I. Mechnikov
Locations (16):
- Russia (16):
  - The First City Clinical Hospital. n.a. E. E. Volosevich, Arkhangelsk
  - Kuzbass Clinical Emergency Hospital named after M.A. Podgorbunsky, Kemerovo
  - Regional clinical hospital №2, Krasnodar
  - Kuban State Medical University, Krasnodar
  - Krasnodar regional hospital №2 (Kuban State Medical University), Krasnodar
  - Regional clinical hospital, Krasnoyarsk
  - Federal research and clinical center of intensive care medicine and rehabilitology, Moscow
  - Loginov Moscow Clinical Scientific Center, Moscow
  - Military Medical Academy, Moscow
  - Moscow cancer research Institute named after P. A. Herzen, Moscow
  - Moscow Regional Research and Clinical Institute, Moscow, Russia, Moscow
  - Moscow regional research clinical Institute named after M. F. Vladimirsky, Moscow
  - Orenburg City N.I. Pirogov Clinical Hospital, Orenburg
  - North-Western State Medical University named after Ilya I. Mechnikov,, Saint Petersburg
  - Regional clinical hospital №2, Vladivostok
  - Clinical city hospital № 40, Yekaterinburg